CLINICAL TRIAL: NCT01080235
Title: Improving Quality of Care for Elderly Patients in the Educational Setting: A Multicenter Exploratory Study of Quality Improvement
Brief Title: Improving Quality of Care for Elderly Patients in the Educational Setting
Acronym: MacyCoVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American Board of Internal Medicine (Other)
Collaborators: The Josiah Macy, Jr. Foundation (Unknown)
Responsible Party: Eric S. Holmboe, MD Senior Vice President for Quality Research and Academic Affairs, American Board of Internal Medicine
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CPS 485
Record Dates: First submitted 2010-03-01; First posted 2010-03-04 (Estimated); Last update posted 2010-03-04 (Estimated); Status verified 2010-03

CONDITIONS: Elderly
Keywords: quality improvement; geriatric care; residency training
MeSH Terms: interventions — Aging

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Control. Forty-two residency programs randomly assigned and stratified according to size, affiliation, geographic location, and presence of geriatrics fellowship. Twenty-one in the control arm. This group will use PIM as a data collection tool during baseline and follow-up time (i.e. audit of 50-75 charts, survey from 50-75 patients, and one system survey). They will not see the summary results of the data collected; they will not be required to complete a quality improvement plan based on the summary data. Local researchers will collect the data. Individual trainees will not do data collection or audits. At both baseline and follow-up, trainees will complete pre and post test surveys of 1) geriatric and 2) quality improvement knowledge, skills, and attitudes.
  Interventions: Other: Geriatric and Quality Improvement toolkit
- 2 (Other): There are 21 residency programs in intervention arm who will 1) use PIM as a data collection tool (local researchers will audit 50-75 charts, survey 50-75 patients, and complete one system survey); 2) Each trainee will audit of up to five patient charts; collect 5 patient surveys; and complete the system survey as a group; 3) Summary data from these data streams will be reviewed by group; then they will design and implement a quality improvement plan; 4) At follow-up, local researchers will re-audit same 50-75 charts, collect surveys from same 50-75 patients, and complete one system survey. At baseline and follow-up, trainees and faculty will complete surveys of geriatric and quality improvement knowledge, skills, and attitudes.
  Interventions: Other: ABIM Care of Vulnerable Elderly Practice Improvement Module; Other: Geriatric and Quality Improvement toolkit

INTERVENTIONS:
Other: ABIM Care of Vulnerable Elderly Practice Improvement Module — The ABIM CoVE PIM is a practice-performance self-evaluation instrument. It is a web-based tool based on nationally recognized guidelines that uses chart abstraction, patient surveys, and a practice system survey in order to generate a performance report focused on a key aspects of care for vulnerable elderly.
  Other Names: Quality improvement module; Practice improvemnet module; Self-assesment in pratice based learning and improvement; PIM in residency
  Arms: 2
Other: Geriatric and Quality Improvement toolkit — A resource toolkit about geriatrics and quality improvement was given to both study arms.
  Other Names: The Improvement Guide by Langley and Nolan; Geriatrics at Your Fingertips; ACOVE Physician Education Program DVD; Online resources; Membership to AGS teaching slides website

SUMMARY:
This is a multi-center exploratory study (each site got local IRB approval) of the impact of an educational toolkit combined with a practice-performance self-evaluation instrument (ABIM Care of the Vulnerable Elderly Practice Improvement Module) on trainee knowledge, skills, and attitudes about practice-based learning and improvement and systems-based practice in the care of elderly patients.

DETAILED DESCRIPTION:
This is a longitudinal quasi-experimental study. Programs will be randomly assigned to either the comparison or intervention group, stratified based on program size, affiliation, geographic location, and presence of a geriatrics fellowship program.

Faculty will be trained in use of the CoVE PIM and in the development and implementation of a quality improvement plan. Residents in the intervention group will perform the medical record audit portion of the CoVE PIM. Patient surveys will be distributed by the residency clinics. The goal will be to audit the medical records of patients who complete the patient survey. Residents in intervention groups will participate in completing the practice system survey as a group. Finally, the residents in the intervention group will use the data from the medical record audit, patient survey, and practice system survey, working with faculty, to develop a quality improvement project to improve care for their geriatric patients.

Local medical record abstractors will be trained to perform a separate medical record audit of a random sample of the same patients identified by the residents for both the intervention and comparison groups. The abstractors will perform both a baseline and follow-up audit and will target the same patients who are still living from the baseline period. The follow-up audit will occur 12 months after completion of the initial PIM data collection phase, or approximately 18 months after the initiation of the study.

Evaluation of study outcomes will occur on the program, resident, and patient level.

ELIGIBILITY:
Inclusion Criteria:

* All residents at a resident clinic site
* Preceptors that are selected by the Champion for a particular resident clinic site
* Patients age 65 years or older for whom any of the following measures would be appropriate: falls prevention, identifying urinary incontinence, screening for depression and cognitive impairment, and providing other preventive care.
* Patients who have been in the practice for at least one year
* Patients who are ambulatory
* Patients who have been seen at least once by the practice within the past 12 months.

Exclusion Criteria:

* Patients under age 65
* Patients who have a terminal illness
* Patients with a life expectancy of less than one-year

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-10; Primary Completion 2007-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Practice Improvement Module (PIM) quality impact | 2 years
  Assess the impact of the Care of the Vulnerable Elderly (CoVE) Practice Improvement Module to improve the quality of care received by elderly patients in the residency ambulatory setting.

SECONDARY OUTCOMES:
Assess satisfaction | 2 years
  Assess resident and faculty satisfaction with the Care of the Vulnerable Elderly Practice Improvement Module.
Assess feasibility | 2 years
  Assess the feasibility of conducting surveys of elderly patients in the residency training setting.
Assess use of geriatric and quality improvement toolkit | 2 years
  Assess the use and impact of an educational toolkit for teaching geriatric quality of care. The analysis will specifically focus on what components of the toolkit are used by programs.
Assess effects of disparities on elder care | 2 years
  Assess the effects of health disparities on the care of elderly patients in a training setting.
Assess barriers in training setting | 2 years
  Assess structural barriers to providing quality care for vulnerable elderly in diverse training settings
Practice Improvement Module impact for knowledge, skills, and attitudes | 2 years
  Assess the impact of the Care of the Vulnerable Elderly Practice Improvement Module to improve the knowledge, skills, and attitudes of residents in the care of specific geriatric conditions.
Practice Improvement Module impact vs traditional | 2 years
  Assess the impact of the Care of the Vulnerable Elderly Practice Improvement Module compared to a traditional educational intervention on residents' knowledge of and attitudes about practice-based learning and improvement, systems based practice, and geriatric care guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Eric S Holmboe, MD, Principal Investigator — American Board of Internal Medicine

REFERENCES:
- See also: ABIM website. Please go to "Helpful Resources" under "Residency Training" to see more information about the CoVE PIM. — http://www.abim.org/